CLINICAL TRIAL: NCT00441636
Title: Treatment Resistant Depression and Obstructive Sleep Apnea: Effect of Treatment With CPAP on Mood, Anxiety and Quality of Life
Brief Title: Treatment Resistant Depression and Obstructive Sleep Apnea, Effect of Continuous Positive Airway Pressure (CPAP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Ruzica Jokic, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSIY-247-06
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Depression; Sleep Apnea, Obstructive
Keywords: depression; CPAP; obstructive sleep apnea
MeSH Terms: conditions — Depression; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CPAP treatment (Experimental): Continuous Positive Airway Pressure (CPAP)for 4 weeks
  Interventions: Device: continuous positive airway pressure (CPAP)
- No CPAP (No Intervention): routine psychiatric care for 4 weeks followed by CPAP titration and initiation after followup measures.
- Control group (No Intervention): No obstructive sleep apnea detected.

INTERVENTIONS:
Device: continuous positive airway pressure (CPAP) — CPAP (Respironics: RemStar plus M-series) machines for treatment of obstructive sleep apnea training for participant required by registered sleep technologist
  Other Names: CPAP - Respironics: RemStar plus M-series
  Arms: CPAP treatment

SUMMARY:
The purpose of the study is to determine the effect on mood and anxiety symptoms of adding CPAP to the psychiatric treatment of patients with TRD (treatment resistant depression) and associated OSA (obstructive sleep apnea).

DETAILED DESCRIPTION:
Primary objective:

What is the effect on mood and anxiety symptoms of adding CPAP to the psychiatric treatment of patients with TRD and associated OSA?

Secondary objectives:

1. How common is co-morbid OSA in patients with treatment resistant unipolar depression referred to a tertiary Mood Disorders Clinic?
2. Is there a difference in daytime functioning (severity of depressive and anxiety symptoms, cognitive function, daytime sleepiness) and sleep quality between patients with TRD diagnosed with OSA compared with patients with TRD who have no OSA?
3. What is the association between sleep fragmentation and hypoxemia and the severity of depression in patients with TRD?

ELIGIBILITY:
Inclusion Criteria:

* Patients with TRD.
* Males and females between the ages of 18 and 65 years who agree to take part and sign the Informed Consent will be invited to participate in the study.
* Patients with co-morbid Dysthymic Disorder, Generalized Anxiety Disorder or Social Anxiety Disorder may be included in the study.

Exclusion Criteria:

* Patients with uncontrolled medical illnesses will not be permitted to participate.
* Patients with a history of current or Bipolar Disorder, Schizophrenia, Panic Disorder, Obsessive-Compulsive Disorder or Anorexia Nervosa.
* Head injury patients resulting in loss of consciousness for more than 10 minutes.
* Patients with epilepsy or severe personality disorders who, at the judgment of the investigators, are not appropriate candidates for the study, will be excluded.
* Patients who do not have the mental or physical capacity to apply the CPAP interface and to plug in and switch on an auto CPAP unit at home will be excluded.
* Blind and/or deaf patients will be excluded.
* Patients who initially decline an offer of CPAP treatment for OSA, and those who prefer conservative treatment options (weight loss, avoidance of alcohol and sedatives) will be excluded.
* Patients with severe claustrophobia, who cannot tolerate any CPAP interface, will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | baseline and 6 weeks

SECONDARY OUTCOMES:
Symbol digit modalities | baseline and 6 weeks
Stroop Test | baseline and 6 weeks
Trail-Making test | baseline and 6 weeks
Pittsburgh Sleep Quality Index (PSQI) | baseline and 6 weeks
Epworth Sleepiness Score (ESS) | baseline and 6 weeks
Beck Anxiety Inventory (BAI) | baseline and 6 weeks
SF-36 questionnaire | baseline and 6 weeks
Profile of mood state (POMS) | baseline and 6 weeks
HAM-D21 | baseline and 6 weeks
  Hamilton depression inventory

CONTACTS AND LOCATIONS:
Overall Officials: Ruzica Jokic, MD, Principal Investigator — Queen's University
Locations (1):
- Providence Continuing Care Centre, Mental Health Services, Kingston, Ontario, Canada